CLINICAL TRIAL: NCT03451370
Title: First-line Combination of Capecitabine and Oxaliplatin + Bevacizumab in Elderly Patients With Metastatic Colorectal Cancer
Brief Title: First-line Combination of Capecitabine and Oxaliplatin Plus Bevacizumab in Elderly Patients With Metastatic Colorectal Cancer
Acronym: COBRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: COBRA
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Elderly Metastatic Colorectal Cancer Patients
Keywords: Bevacizumab; Capecitabine; Oxaliplatin; CRASH score; ECOG PS; G8 score
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Capecitabine — 750 mg/sqm/bid, day 2 to 15; if toxicities grade ≥2 do not occur, pts may subsequently receive capecitabine 1000 mg/sqm/bid, day 2 to 15 starting the second cycle based on investigator's choice.
  To be repeated every 3 weeks (21 days), for a maximum of 8 cycles.
  If no progression occurs, pts will receive maintenance capecitabine (starting at the same dose used at the last cycle of the induction treatment) plus bevacizumab every 3 weeks (21 days), until disease progression, unacceptable toxicity or patient's refusal.
Drug: Oxaliplatin — 100 mg/sqm iv over 2 hours, day 1 To be repeated every 3 weeks (21 days), for a maximum of 8 cycles.
Drug: Bevacizumab — 7.5 mg/kg iv over 90 minutes, day 1; if the first infusion is tolerated, then subsequent infusions may be administered in 30 minutes.
  If no progression occurs, pts will receive maintenance capecitabine (starting at the same dose used at the last cycle of the induction treatment) plus bevacizumab every 3 weeks (21 days), until disease progression, unacceptable toxicity or patient's refusal. To be repeated every 3 weeks (21 days), for a maximum of 8 cycles.

SUMMARY:
* Oxaliplatin-based doublets plus bevacizumab are standard first-line therapy options for patients (pts) with metastatic colorectal cancer (mCRC). Slight adjustments in chemo-dosage are commonly applied in routinely practice to elderly pts, but those modified schedules have never been standardized
* The addition of oxaliplatin versus no oxaliplatin to treatment with 5-fluorouracil in older and frail untreated pts with mCRC resulted in a non-statistically significant trend toward improvement in Progression Free Survival (PFS) and a lack of benefit in Overall Survival (OS)
* In elderly pts deemed unfit for an upfront combined chemotherapy a fluoropyrimide-based monotherapy plus bevacizumab is considered a reasonable first-line treatment
* Clinical definition of elderly (over 70 years old) pts with CRC that may deserve a more or less intensive combination therapy is still debated. The cut-off of 75 years old combined with ECOG PS assessment is a reasonable approach for clearly defining candidates to different approaches
* Several geriatric screening tools have been used to identify pts with a geriatric profile potentially predicting for overall survival and risk of toxicity. The G8 screening tool has been already validated in pts with cancer showing the strongest prognostic value for OS; the CRASH score is able to stratify pts according an estimated risk of treatment-related toxicities

On the basis of these considerations, we designed the present observational study of first-line therapy with bevacizumab in combination with capecitabine and oxaliplatin in previously untreated elderly pts affected by unresectable mCRC in order to evaluate its efficacy in real world practice (as measured by progression free survival)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal cancer.
* Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
* Indication to oxaliplatin, capecitabine and bevacizumab as first line treatment.
* At least one measurable lesion according to RECIST1.1 criteria.
* Availability of a tumoral sample (primary and/or metastatic sites).
* Age ≥ 70 years.
* ECOG PS (Eastern Cooperative Oncology Group - Performance Status) 1 or 2 for pts aged 70 to 75 years; ECOG PS 0 or 1 for pts aged > 75 years.
* Life expectancy of at least 12 weeks.
* Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse.
* Laboratory Requirements:

  * Neutrophils ≥1.5 x 109/L,
  * Platelets ≥100 x 109/L,
  * Hgb ≥ 9 g/dl.
  * Total bilirubin ≤ 1.5 time the upper-normal limits (UNL) of the normal values and ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases),
  * Alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases),
  * Creatinine clearance ≥ 50 mL/min or serum creatinine ≤1.5 x UNL,
  * Urine dipstick of proteinuria <2+. Pts discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate <1 g of protein/24 hr.
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception as approved by the investigator (i.e. barrier contraceptive measure or oral contraception, total abstinence) during the study and until 6 months after the last treatment.
* Geriatric assessment by means of G8 screening tool and CRASH score.
* Written informed consent to study procedures and to molecular analyses before pts registration.
* Will and ability to comply with the protocol.

Exclusion Criteria:

criteria

* Previous adjuvant oxaliplatin-containing chemotherapy.
* Previous treatment with bevacizumab.
* Previous systemic treatment for the metastatic disease.
* Previous radiotherapy treatment to any site within 4 weeks before the study.
* Evidence of untreated brain metastases or spinal cord compression or primary brain tumours.
* History or evidence upon physical examination of CNS disease unless adequately treated.
* Symptomatic peripheral neuropathy > 1 grade NCIC-CTG criteria.
* Serious, non-healing wound, ulcer, or bone fracture.
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication.
* Any previous venous thromboembolism > NCI CTCAE Grade 3.
* History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
* Current ongoing treatment with anticoagulants for therapeutic purposes.
* Chronic, daily treatment with high-dose aspirin (>325 mg/day).
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration or putting the patient at high risk for treatment-related toxicities.
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Contraindications for the use of corticosteroids and antihistamines as premedication or known hypersensitivity to any other component of the study drugs.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly (> 70 years) patients with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 28 months
  PFS is defined as the time from study enrollment to the first documentation of objective disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy